CLINICAL TRIAL: NCT05621694
Title: Exploring Oxytocin Response to Meditative Movement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arizona State University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00006571
Record Dates: First submitted 2022-05-25; First posted 2022-11-18 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2023-09

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Tai Ji

STUDY DESIGN:
Intervention Model Description: Meditative movement practice: Tai Chi Easy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Qigong/Tai Chi Intervention (Experimental): Tai chi and Qigong combined into a simplified, standard practice, "Tai Chi Easy"
  Interventions: Behavioral: Tai Chi Easy

INTERVENTIONS:
Behavioral: Tai Chi Easy — A meditative movement practice that includes simple qigong movement/breath practices and single, repeated tai chi movements taught to generate a meditative state and flow
  Other Names: Qigong/Tai Chi; taiji

SUMMARY:
This pilot study is designed to test effects of a single session of meditative movement (Tai Chi Easy) on older adults' blood pressure, perceptions of connection, mood, and oxytocin levels.

DETAILED DESCRIPTION:
Endogenous oxytocin (the "cuddle hormone") is associated with lowering blood pressure (BP), suggesting that finding ways to increase oxytocin even in the absence of social connection, may be beneficial. Meditative movement emphasizing breath, meditative state and flow-inducing movements holds potential for reducing BP, improving mood and releasing oxytocin. In a single-group pilot study we exposed 21 OAs with mild-moderate hypertension to a 50-minute "Tai Chi Easy (TCE)" (simplified Tai Chi/Qigong) session, collecting BP, saliva samples for oxytocin, and psychosocial measures (connection, mood) pre/post intervention.

ELIGIBILITY:
Inclusion Criteria:

* Age 55-80 --BP above 120/80 -

Exclusion Criteria:

* having a neurologic disorder such as Parkinson's, seizure disorder, multiple sclerosis, Alzheimer's disease
* answered "yes" to one or more questions on the Physical Activity Readiness Questionnaire (PAR-Q). The PAR-Q is a seven-question assessment that determines one's readiness, safety and ability to engage in physical activity and is safely validated for older adults

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2017-09-30 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Change in Blood Pressure | Change from baseline (pre-intervention) blood pressure to immediately after the 50-minute intervention
  Using blood pressure cuff, conducting two consecutive readings of systolic and diastolic

SECONDARY OUTCOMES:
Change in Profile of Mood States; Short Form | Change from pre-intervention mood to immediately post-50-minute intervention point
  Using only subscales for depression and tension, 14 items with response format 0-4, reporting mean of responses, range 0-4 with higher scores indicating higher levels of depression and tension.
Change in perception of Connection (this is not a published scale, no formal name, created for this study) | Change from pre-intervention to immediately after the 50-minute intervention
  Two items assessing perception of connection with others and connection with self, score range
Change in Salivary Oxytocin | Change from pre-intervention to immediately after the 50-minute intervention
  Saliva collection pre and post-intervention

OTHER OUTCOMES:
The De Jong Gierveld Loneliness Scale | pre-intervention only
  6 items each scored either 0 (not at all) 1 (somewhat lonely) or 2 (more lonely), score is computed as a mean across items, range 0-6 with higher scores indicating more loneliness
Flow State Scale | immediately after the intervention
  Used to assess perceptions of the experience of flow while performing the Tai Chi Easy intervention. 36 items, Score range 36-80, high scores indicate greater sense of flow.
Meditative Movement Inventory | immediately after the intervention
  Scales that assess the experience of meditative state and breath focus during intervention, 11 items, score range 11-66 (or reported as a mean of the scores on the scale, then 1-6 range), with higher numbers indicating less breath focus and meditative state.

CONTACTS AND LOCATIONS:
Overall Officials: Linda K Larkey, PhD, Principal Investigator — Arizona State University
Locations (2):
- United States (2):
  - Arizona State University Downtown Campus, Phoenix, Arizona
  - Arizona State University, Phoenix, Arizona

IPD SHARING:
Plan to Share IPD: Yes
Will publish with indication that IPD data that is de-identified is available upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available after study results are published and for 5 years after.
Access Criteria: Requests from active researchers with current positions in research institutions will be reviewed by PI

REFERENCES:
- [Result] Larkey LK, James T, Han S, James DL. Pilot study of Qigong/Tai Chi Easy acute effects of meditative movement, breath focus and "flow" on blood pressure, mood and oxytocin in older adults. Complement Ther Med. 2023 Mar;72:102918. doi: 10.1016/j.ctim.2023.102918. Epub 2023 Jan 7. PMID 36626941